CLINICAL TRIAL: NCT04274374
Title: Impact of a Gluten-free Diet on Quality of Life in Patients With Axial Spondyloarthritis: Study Protocol of a Randomized Double-blind Placebo-controlled Trial
Brief Title: Impact of a Gluten-free Diet on Quality of Life in Patients With Axial Spondyloarthritis.
Acronym: GlutenSPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: PANZANI (Unknown); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC IR 2017 COUDERC; 2018-A00309-46 (Other: ANSM)
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Ankylosing Spondyloarthritis
Keywords: spondyloarthritis; ankylosing spondylitis; gluten-free diet; gut microbiota
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): In the experimental arm will receive at least 6 gluten-free breads per day + 200 g of gluten-free penne pasta per week + 6 rice flavor capsules per day
  Interventions: Dietary Supplement: Gluten-Free Diet
- control arm (Active Comparator): the control arm will received 6 gluten-containing breads per day + 200 g of gluten-containing penne pasta per week + 6 vital gluten-containing capsules per day
  Interventions: Dietary Supplement: Gluten Diet

INTERVENTIONS:
Dietary Supplement: Gluten-Free Diet — Dietary supplement without gluten
  Arms: experimental arm
Dietary Supplement: Gluten Diet — Dietary supplement with gluten
  Arms: control arm

SUMMARY:
Subclinical intestinal inflammation and gut dysbiosis have been reported in patients with spondyloarthritis (SpA). In common practice, rheumatologists are increasingly confronted with patients with inflammatory rheumatism who are on gluten-free diets (GFDs), despite the lack of reliable data from controlled studies. This study aims to determine the impact of a GFD on the quality of life of patients with axial SpA.

DETAILED DESCRIPTION:
The GlutenSpA study is a 24-week, randomized, double-blinded, placebo-controlled, multicenter trial. Patients with axial SpA (n=200) will follow a 16-week GFD and be randomly assigned (1:1) to an experimental or control arm. In the experimental arm with receive at least 6 gluten-free breads per day + 200 g of gluten-free penne pasta per week + 6 rice flavor capsules per day. The control arm will receive at least 6 gluten-containing breads per day + 200 g of gluten-containing penne pasta per week + 6 vital gluten-containing capsules per day.

At baseline, the dietician will explain to the patients how to properly follow a GFD during a face-to-face interview. The patient's compliance to the GFD will be evaluated by the dietician at S2, S16, an S24 using an online 3-day alimentary questionnaire.

The bread and penne pasta were chosen for their visual resemblance and similar taste to maximize the blindness of the study. In order to reach the daily amount of gluten in a standard diet (estimated in France between 10 and 15 g/d) in the control arm, each day patients will have to ingest six capsules of vital gluten wheat made for the study. Vital gluten flour is an over-the-counter food supplement used to enrich a protein diet or as a base for making products, such as seitan. Capsules will be made using commercially available vital gluten and contain 0.35 g of gluten per capsule. The total amount of gluten in the control arm will be approximately 10.5 g/day.

After the 16-week GFD, patients will be offered to follow or not follow the GFD according to their own decision for an 8-week open-labelled follow-up period. The study duration for each patient is 24 weeks. The patient recruitment is expected to last 2 years

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of axial SpA defined by ASAS criteria
* Rheumatologist not wish to change the treatment within 4 months of inclusion,
* stable treatment (NSAID and/or DMARD) for at least 3 months but no corticosteroid infiltration in the month prior to inclusion,
* able to follow a GFD and to provide written informed consent and submit to the requirements of the study

Exclusion Criteria:

* Any diet at the time of inclusion or within 3 months prior to inclusion;
* have a history of celiac disease;
* received antibiotic treatment within 3 months of inclusion or are taking a probiotic;
* are pregnant, breastfeeding,
* not covered by social security;
* minors or adults under the protection of the law or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the variation in quality of life evaluated variation inby the Assessment of SpondyloArthritis international Society (ASAS) Health Index | Change from baseline ASAS HI score at 16 weeks
  The self-report questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EF) in patients with SpA. The total sum of the ASAS HI ranges from 0-17, with a lower score indicating a better health status.

SECONDARY OUTCOMES:
effects of a 16-week GFD versus placebo diet on the activity of SpA evaluated by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). | Change from baseline BASDAI score at 16 weeks
  The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. Scores of 4 or greater suggest suboptimal control of disease,
effects of a 16-week GFD versus placebo diet on parameters of inflammation evaluated by the erythrocyte sedimentation rate (ESR). | Change from baseline ESR at 16 weeks
  An ESR is a type of blood test that measures how quickly erythrocytes settle at the bottom of a test tube that contains a blood sample. Normally, red blood cells settle relatively slowly. A faster-than-normal rate may indicate inflammation in the body.
effects of a 16-week GFD versus placebo diet on parameters of inflammation evaluated by the C-reactive protein (CRP) | Change from baseline CRP at 16 weeks
  A c-reactive protein test measures the level of c-reactive protein (CRP) in your blood. CRP is a protein made by your liver. It's sent into your bloodstream in response to inflammation. Normally, you have low levels of c-reactive protein in your blood. High levels may be sign of a serious infection or other disorder.
effects of a 16-week GFD versus placebo diet on fatigue assessed by the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale. | Change from baseline FACIT score at 16 weeks
  The FACIT Fatigue Scale is a short, 13-item, that measures an individual's level of fatigue during their usual daily activities over the past week. Score range 0-52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life
effects of a 16-week GFD versus placebo diet on depression evaluated by the Hospital anxiety and depression scale (HAD) | Change from baseline HAD score at 16 weeks
  The HAD scale is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. cut-off point of 8/21 for anxiety or depression
Variations in the abundance and type of different bacterial species found in the intestinal microbiota for a subgroup of patients | Change from baseline abundance and types of bacteria at 16 weeks
  The microbiota will be analyzed in a subgroup of patients (n = 40) using stool samples collected at J0 and S16
effects of a 16-week GFD versus placebo diet on functional disability asssessed by Bath Ankylosing Spondylitis Functionnal Index (BASFI) questionnaire | Change from baseline BASFI score at 16 weeks and at 24 weeks
  Functional disability index consisting of 10 questions. The final score is calculated on 100 points. The higher the score, the greater the handicap.
effects of a 16-week GFD versus placebo diet on the persistence of fibromyalgia syndrome | Persistence of fibromyalgia syndrome at week 16 and 24 (if present at inclusion)
  the Fibromyalgia rapid screening tool (FIRST) questionnaire makes it possible to screen for fibromyalgia syndrome quickly and easily. The FIRST questionnaire consists of 6 questions. A score of 5/6 or higher indicates definite fibromyalgia syndrome
Evaluation of compliance with the GFD by an interview with the dietician | at week 16
  The patient's compliance to the GFD will be evaluated by the dietician using an online 3-day alimentary questionnaire. The patient will have to postpone all food consumed and its quantity during the last 3 days before the consultation with the dietician
effects of a 16-week GFD versus placebo diet on body mass index (BMI) | Change from baseline BMI at week 16 and 24
  The BMI will be calculated by the formula (height/weight²).
effects of a 16-week GFD versus placebo diet on Homeostasis Model Assessment of insulin resistance (HOMA-IR) | Change from baseline insulin resistance at week 16
  Insulin resistance will be calculated by the following formula : fasting blood glucose (mmol / l) x fasting insulin (μmol/l) /22.5. A score greater than or equal to 3 indicates insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Marion Couderc, MD, Principal Investigator — CHU de Clermont-Ferrand
Locations (7):
- France (7):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - Assistance Publique - Hôpitaux de Paris (AP-HP) - Hôpital Cochin, Paris
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couderc M, Pereira B, Schaeverbeke T, Thomas T, Chapurlat R, Gaudin P, Morel J, Dougados M, Soubrier M. GlutenSpA trial: protocol for a randomised double-blind placebo-controlled trial of the impact of a gluten-free diet on quality of life in patients with axial spondyloarthritis. BMJ Open. 2020 Nov 20;10(11):e038715. doi: 10.1136/bmjopen-2020-038715. PMID 33444189